CLINICAL TRIAL: NCT04389476
Title: The Impact and Coping Strategy of Taiwan Society and Medical and Nursing Institutes Toward the Biological Disaster-- Corona Virus Disease 2019 (COVID-19) as An Example
Brief Title: The Impact and Coping Strategy of COVID-19 Among Taiwan Society and Medical and Nursing Institutes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Kai-Suan Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Frank Huang-Chih Chou, MD, MS, PhD, President, Kaohsiung Municipal Kai-Suan Psychiatric Hospital, Kaohsiung Kai-Suan Psychiatric Hospital
Other Study IDs: KSPH-2020-03
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: The Psychological Impact of COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Medical staff in high contact with patients
  Interventions: Other: Standardized crisis management and coping protocol plan toward Coronavirus disease 2019 (COVID-19)
- Other personnel in low contact with patients
  Interventions: Other: Standardized crisis management and coping protocol plan toward Coronavirus disease 2019 (COVID-19)
- Patients
  Interventions: Other: Standardized crisis management and coping protocol plan toward Coronavirus disease 2019 (COVID-19)
- Community residents
  Interventions: Other: Standardized crisis management and coping protocol plan toward Coronavirus disease 2019 (COVID-19)

INTERVENTIONS:
Other: Standardized crisis management and coping protocol plan toward Coronavirus disease 2019 (COVID-19) — Establish standardized crisis management and coping protocol plan toward Coronavirus disease 2019 (COVID-19) for the different tiers of medical staff, patients, and community residents.
  Then explore the psychological impact and mental disabilities under the intervention and controlling related factors.

SUMMARY:
The Coronavirus disease 2019 (COVID-19) had its outbreak in late 2019 in China and is considered a biological disaster. With medical organizations and staff on the frontline, the investigators should conduct assessments, for the different tiers of medical staff, patients, and community residents, on the short- term psychological and mental disabilities or danger factors that they might have faced. As such, the investigators can design and establish a set of evaluative indicators of the risks of biological disasters, and strategies to manage guide and cope, and internal/ external testing strategies. These work in guaranteeing quality and performance, and as such, establishing "Digital Platform for Integrated Research of Coronavirus disease 2019 (COVID-19)".

ELIGIBILITY:
Inclusion Criteria:

* 1.>20 years old. 2. Medical staff and patients from different tiers hospitals in Taiwan. 3.Community residents in Taiwan

Exclusion Criteria:

* 1.< 20 years old. 2. These cases who had disabilities can't complete our assessments.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Medical staff in high contact with patients 2. Other personnel in low contact with patients 3. Patients 4. Community residents.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Psychological impacts by CoronaVirus Disease 2019(COVID-19) | 3 years
  Acute and chronic psychological impacts on medical and nursing staff and the mass public by CoronaVirus Disease 2019(COVID-19)

IPD SHARING:
Plan to Share IPD: Undecided